CLINICAL TRIAL: NCT05531994
Title: Bioequivalence Study of Montelukast Sodium Oral Thin Film and Chewable Tablet in Fed Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: QL-XZ1-013-02
Record Dates: First submitted 2022-09-04; First posted 2022-09-08 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Water

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TR (Other): Administration order: montelukast sodium oral thin films with water, montelukast sodium chewable tablets with water.
  Interventions: Drug: Montelukast sodium oral thin films with water (T); Drug: Montelukast sodium chewable tablets with water (R)
- RT (Other): Administration order: montelukast sodium chewable tablets with water, montelukast sodium oral thin films with water.
  Interventions: Drug: Montelukast sodium oral thin films with water (T); Drug: Montelukast sodium chewable tablets with water (R)

INTERVENTIONS:
Drug: Montelukast sodium oral thin films with water (T) — Single-dose montelukast sodium oral thin film 5mg under fed condition with water 240 mL
Drug: Montelukast sodium chewable tablets with water (R) — Single-dose montelukast sodium chewable tablet 5mg under fed condition with water 240 mL

SUMMARY:
This study aimed to evaluate the pharmacokinetic characteristics of montelukast sodium oral thin films and the bioequivalence between oral thin films and chewable tablets in healthy chinese volunteers under fed condition.

ELIGIBILITY:
Inclusion Criteria:

* Fully understood and voluntarily signed the informed consent form
* With high compliance
* BMI 18.6-28.5 kg/m^2, and with weight ≥ 50 kg for male, or ≥ 45 kg for female

Exclusion Criteria:

* Allergic to any component of study drugs, other leukotriene receptor antagonists, sulfonamides, or non-steroidal anti-inflammatory drugs
* With clinically relevantly abnormal vital sign, examination, or clinically relevant disease
* Had drug abuse within 3 months before screening or positive in drug of abuse test
* With any routine use of drugs
* Received major surgery within 6 months before study drug administration or planned to receive major surgery during study period
* With average number of cigarettes smoked > 5/day within 3 months before screening or refused to suspend smoking from 24 hours before study drug administration throughout study period
* With average alcohol consumption > 14 units/week within 6 months before screening or refused to suspend alcohol consumption from 24 hours before study drug administration throughout study period
* With average tea, coffee, or other drink with caffeine consumption > 8*250 mL/day, or refused to suspend tea, coffee, other drink with caffeine, or grape fruit juice consumption from 24 hours before study drug administration throughout study period
* Lost or donated blood > 200 mL within 3 months, or donated platelet > 24 U within 1 months before study drug administration
* Received any drug within 14 days before study drug administration
* Received any drug of other clinical trial within 3 months before study drug administration
* Received any vaccine within 4 weeks before study drug administration
* Planned for pregnancy within 3 months after informed consent form signed or refused to use adequate contraception (excluding contraceptive drug)
* For female, pregnant, breastfeeding, received oral contraceptives within 30 days, or contraceptive injection or implant within 6 months before study drug administration
* For pregnancy-capable female, had unprotected sexual contact within 14 days before study drug administration

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-11-27 (Actual); Primary Completion 2019-05-14 (Actual); Study Completion 2019-05-14 (Actual)

PRIMARY OUTCOMES:
Cmax | 0-24 hours
  The maximum plasma drug concentration
AUC0-t | 0-24 hours
  The area under the concentration-time curve from dosing to time t
AUC0-∞ | 0-24 hours
  The area under the concentration-time curve extrapolated to infinity

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoai He, Principal Investigator — Haikou People's Hospital
Locations (1):
- Haikou People's Hospital, Haikou, Hainan, China

REFERENCES:
- [Derived] Zhu G, Wang L, Han S, Peng H, Tong M, Gu X, Hu H, Wang Y, Lv Z, He X. Pharmacokinetics and bioequivalence study of montelukast sodium oral soluble film and chewable tablet in healthy Chinese volunteers: randomized trials under fasting and fed conditions. Ann Transl Med. 2023 Jan 31;11(2):93. doi: 10.21037/atm-22-6485. PMID 36819512